CLINICAL TRIAL: NCT04926831
Title: Phase II Trial of Neoadjuvant and Adjuvant Capmatinib in Participants With Stages IB-IIIA, N2 and Selected IIIB (T3N2 or T4N2) NSCLC With MET Exon 14 Skipping Mutation or High MET Amplification (Geometry-N)
Brief Title: Phase II of Neoadjuvant and Adjuvant Capmatinib in NSCLC
Acronym: Geometry-N
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to recruitment challenges.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280AUS12
Record Dates: First submitted 2021-06-14; First posted 2021-06-15 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Mesenchymal Epithelial Transition (MET); MET exon 14 skipping mutation; High MET amplification; Neoadjuvant; Prior to surgery; Adjuvant; After surgery; INC280; MET inhibition; adult; capmatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — capmatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (MET exon 14 skipping mutations) (Experimental): The study treatment started on Cycle 1 Day 1 with the first administration of capmatinib 400 mg twice a day (b.i.d.). The participants were planned to receive study treatment for a maximum of 3 years following surgery or until early discontinuation.
  Interventions: Drug: capmatinib
- Cohort B (high MET amplification) (Experimental): The study treatment started on Cycle 1 Day 1 with the first administration of capmatinib 400 mg twice a day (b.i.d.). The participants were planned to receive study treatment for a maximum of 3 years following surgery or until early discontinuation.
  Interventions: Drug: capmatinib

INTERVENTIONS:
Drug: capmatinib — 150 mg and 200 mg tablets for oral administration
  Other Names: INC280

SUMMARY:
This study was planned to determine if neoadjuvant capmatinib could improve the major pathological response (MPR) in patients with Stage IB-IIIA, N2 and selected IIIB (T3N2 or T4N2) lung cancers with Mesenchymal Epithelial Transition (MET) exon 14 mutations and/or high MET amplification beyond those achieved with surgery, chemotherapy, and radiation. Treatment was to be continued with capmatinib in the adjuvant setting to evaluate the potential clinical benefit of extended therapy.

The purpose of this study is to determine if neoadjuvant capmatinib can improve outcomes in participants with stages I-IIIA non-small cell lung cancer with MET exon 14 mutations and/or high MET amplification beyond those achieved with surgery, chemotherapy, and radiation.

DETAILED DESCRIPTION:
This was a Phase II, two cohort, two stage study of capmatinib given for 8 weeks (2 cycles) prior to surgical resection, followed by three-year capmatinib treatment in adjuvant setting. Surgery had to be performed up to 2 weeks after the last dose of neoadjuvant study treatment.

There were 2 molecularly defined cohorts enrolled in parallel:

* Cohort A: MET exon 14 skipping mutations, irrespective of MET GCN or
* Cohort B: high level MET amplification (MET: GCN ≥ 10 by FISH or FoundationOne CDx NGS using tumor tissue).

Approximately 42 participants were aimed to be enrolled in the study, with 21 participants per cohort. This was planned to obtain 38 evaluable participants, 19 per each cohort. Participants who had both MET exon 14 skipping mutations and high-level MET amplification were planned to be enrolled into Cohort A. An evaluable subject received the neoadjuvant treatment and subsequently underwent surgery, resulting in a pathological response.

The study recruitment was prematurely discontinued due to significant recruitment challenges leading to termination of the study. The challenges included the rarity of the mutation and site initiation delays caused by staff shortages associated with COVID-19. As a result, only 4 subjects were enrolled and treated in Cohort A.

ELIGIBILITY:
Key inclusion criteria:

1. Adult ≥ 18 years of age at the time of informed consent.
2. Histologically confirmed NSCLC Stage IB-IIIA, N2 and selected IIIB (T3N2 or T4N2) (per AJCC 8th edition), deemed suitable for primary resection by treating surgeon (T4 tumors with mediastinal organ invasion were not eligible for enrollment).
3. Participant must have MET exon 14 mutation and/or high-level MET amplification (MET: GCN ≥ 10) as determined by a CLIA certified laboratory. High level MET amplification must be identified by FISH in a CLIA certified laboratory or FoundationOne CDx NGS (other NGS-based methods without adjusting for tumor content % cannot be accepted).
4. Participants must be eligible for surgery and scheduled for surgical resection within approximately 2 weeks after the last dose of neoadjuvant study treatment.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.

Key exclusion criteria:

1. Participants with unresectable or metastatic disease. All participants should have brain imaging (either MRI brain or CT brain with contrast) prior to enrollment to exclude brain metastasis.
2. Presence or history of a malignant disease that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
3. Prior treatment with any MET inhibitor or HGF-targeting therapy.
4. Participants with other known oncogenic driver alterations.
5. Prior systemic anti-cancer therapy (chemotherapy, immunotherapy, biologic therapy, vaccine) or investigational agents for NSCLC.
6. Participants with known hypersensitivity to capmatinib and any of the excipients of capmatinib (crospovidone, mannitol, microcrystalline cellulose, povidone, sodium lauryl sulfate, magnesium stearate, colloidal silicon dioxide, and various coating premixes).

Other protocol-defined inclusion/exclusion criteria may apply at the end

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - UCLA Oncology Hematology ., La Jolla, California
  - UCLA Oncology Hematology, La Jolla, California
  - University of California Davis Cancer Center ., Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Fairfax Northern Virginia Hem Onc ., Fairfax, Virginia
  - Fairfax Northern Virginia Hem Onc, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2549

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 3 centers in the USA.
Period: Overall Study
Arm/Group | Cohort A (MET Exon 14 Skipping Mutations)
Started | 4
Completed | 0
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cohort A (MET Exon 14 Skipping Mutations)
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: Years] | 78.25 [74 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Major Pathological Response (MPR) Rate
Description: The primary efficacy variable was MPR rate, defined as the proportion of participants with ≤ 10% residual viable cancer cells. MPR rate was to be assessed via local review for primary analysis. MPR assessment in tumor samples was collected at time of resection.
  Due to low number of participants and limited data, analysis related to the primary endpoint was not performed.
Time Frame: Baseline up to time of surgery (approximately 8 to 10 weeks after first dose)
Population: All enrolled participants with tumor tissue samples
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (MET Exon 14 Skipping Mutations)
Number analyzed (Participants) | 3
Participants
  Responder as per local review | 1
  Responder as per central review | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) was defined as the percentage participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response ( PR) according to RECIST v1.1. BOR was the observed response at the assessment performed prior to surgery via local review.
Time Frame: Baseline up to time of surgery (approximately 8 - 10 weeks after first dose)
Population: All enrolled participants with tumor tissue samples
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (MET Exon 14 Skipping Mutations)
Number analyzed (Participants) | 3
Participants | 1

3. Secondary Outcome: Complete Pathologic Response (pCR) Rate
Description: Complete pathologic response (pCR) rate ws defined as the percentage of participants with no residual viable cancer cells. pCR rate was assessed via both central and local review.
Time Frame: Baseline up to time of surgery (approximately. 8- 10 weeks after first dose)
Population: All enrolled participants with tumor tissue samples
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (MET Exon 14 Skipping Mutations)
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Disease Free Survival (DFS)
Description: Disease Free Survival (DFS) was defined as the time from the date of first adjuvant treatment to the date of the first documented disease recurrence as assessed by local investigator radiologically or death due to any cause. In case of non-conclusive radiological evidence, a biopsy was to be performed to confirm recurrence and used as DFS event. DFS events were assessed locally.
Time Frame: From time of surgery to Months 24, 36, and 60
Population: All enrolled participants. Due to early discontinuation of the study, no participants reached month 24 (no data was collected/analyzed for the endpoint).
Arm/Group | Cohort A (MET Exon 14 Skipping Mutations)
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Adverse Events and Serious Adverse Events as Assessed by CTCAE Criteria
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  Treatment emergent Adverse Event (TEAEs) in this study were events that started after the first dose of study treatment and until 30 days after the last dose of study treatment, or events present prior to the first dose of treatment which increased in severity based on preferred term within 30 days after the last study treatment.
Time Frame: Baseline up to 30 days after last dose of study medication, assessed up to approximately 20 months
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (MET Exon 14 Skipping Mutations)
Number analyzed (Participants) | 4
Participants
  Adverse Events (AEs) | 4
  AEs leading to study treatment discontinuation | 2
  AEs leading to dose adjustment and/or interruption | 4
  Serious Adverse Events (SAEs) | 3
  SAEs related to study treatment | 0
  Fatal SAEs | 1

ADVERSE EVENTS:
Time Frame: On-treatment adverse events and deaths were reported from first dose of study medication up to 30 days after last dose of study medication, assessed up to approximately 20 months.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The safety analysis were done on the safety population, which included all randomized subjects who received at least one dose of study medication.
Arm/Group | Cohort A (MET Exon 14 Skipping Mutations)
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (MET Exon 14 Skipping Mutations) (N=4)
Inguinal hernia (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (MET Exon 14 Skipping Mutations) (N=4)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Sinus arrest (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anorectal discomfort (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 2
Generalised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pain (General disorders) | 1
Physical deconditioning (General disorders) | 1
Pyrexia (General disorders) | 1
Sensation of foreign body (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 2
Escherichia urinary tract infection (Infections and infestations) | 1
Streptococcal urinary tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Incision site erythema (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Fibrin D dimer increased (Investigations) | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1
Troponin T increased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Sleep terror (Psychiatric disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT04926831/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04926831/SAP_001.pdf